CLINICAL TRIAL: NCT00975910
Title: Effect of Lidocaine in Antiarrhythmic Dosage on Postoperative Cognitive Dysfunction in Supratentorial Craniotomy Dysfunction in Supratentorial Craniotomy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Capital Medical University (Other)
Collaborators: State University of New York - Downstate Medical Center (Other)
Responsible Party: Principal Investigator, Wei Zhang, attending, Capital Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 20090801
Record Dates: First submitted 2009-09-11; First posted 2009-09-14 (Estimated); Last update posted 2013-05-22 (Estimated); Status verified 2013-05

CONDITIONS: Supratentorial Craniotomy Dysfunction
Keywords: Supratentorial Craniotomy
MeSH Terms: interventions — Lidocaine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Saline (Placebo Comparator)
  Interventions: Drug: saline
- Lidocaine (Active Comparator)
  Interventions: Drug: lidocaine

INTERVENTIONS:
Drug: lidocaine — Lidocaine arm: lidocaine (2%) as an intravenous bolus (1.5 mg/kg) during induction followed by an intravenous infusion (2 mg. kg(-1).h(-1)) after induction until at the end of surgery
  Arms: Lidocaine
Drug: saline — Saline arm: infused at the same rate as lidocaine
  Arms: Saline

SUMMARY:
The purpose of this study is to investigate the effect of lidocaine in antiarrhythmic dosage on postoperative cognitive dysfunction in supratentorial craniotomy.

ELIGIBILITY:
Inclusion Criteria:

* 18-60 years old, ASA physical status I or II, BMI<30
* Scheduled for elective supratentorial craniotomy
* MMSE<24 before operation
* Cooperative and given informed consent in person

Exclusion Criteria:

* History of mental or psychiatric disorders
* Contraindicated to internal jugular venous catheterization
* Pregnant or lactating female
* History of systemic malignant tumor or diabetes
* Previously treated with this protocol or participated in another study within previous 30 days
* Suspected history of allergic reaction or intolerance to amides or other anesthetic agents in this study
* History of alcohol abuse and/or drug abuse within previous one year
* History or a family history of malignant hyperthermia

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2009-09; Primary Completion 2012-05 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Mini-Mental State Examination (MMSE) | Preoperatively, 3 days and 3 months postoperatively
Montreal Cognitive Assessment (MoCA) | Preoperatively, 3 days and 3 months postoperatively
Hamilton Depression Scale (HAMD) | Preoperatively, 3 days and 3 months postoperatively
Clinical Dementia Rating (CDR) | Preoperatively, 3 days and 3 months postoperatively
Confusion Assessment Method for the Diagnosis of Delirium in the Intensive Care unit (ICU) (CAM-ICU) | 1 day and 3 days postoperatively

SECONDARY OUTCOMES:
AjDO2 (Arterial Jugular Difference) | Injection of test dosage, 1 hour, 2 hours, 3 hours after injection of test dosage, end of surgery
AjDGlc | Injection of test dosage, 1 hour, 2 hours, 3 hours after injection of test dosage, end of surgery
AjDGlutamate | Injection of test dosage, 1 hour, 2 hours, 3 hours after injection of test dosage, end of surgery
AjDLct | Injection of test dosage, 1 hour, 2 hours, 3 hours after injection of test dosage, end of surgery
S100 | Injection of test dosage, end of surgery, 24 hours after operation
Amyloid-β protein(Aβ) | Injection of test dosage, end of surgery, 24 hours after operation

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology,Beijing Tiantan Hospital, Capital Medical University, Beijing, Beijing Municipality, China